CLINICAL TRIAL: NCT00112047
Title: A Phase 3, Randomized, Multicenter Study of the Treatment of Antiretroviral-Naive HIV-1 Infected Subjects Comparing Tenofovir Disoproxil Fumarate and Emtricitabine in Combination With Efavirenz vs Combivir (Lamivudine/Zidovudine) and Efavirenz
Brief Title: Tenofovir Disoproxil Fumarate/Emtricitabine/Efavirenz Versus Combivir/Efavirenz in Antiretroviral-Naive HIV-1 Infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Steven Chuck MD, Vice President, HIV Therapeutics, Clinical Research, Gilead Sciences, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-01-934
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Results first posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Emtricitabine; Racivir; Tenofovir; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EFV+CBV (Active Comparator): Participants in this group received EFV 600 mg once daily + Combivir ([CBV]; the fixed dose combination pill containing lamivudine 150 mg + zidovudine 300 mg) taken twice daily from the start of the study until Week 144. At Week 144 all participants who opted to roll over into the additional 96-week study extension received Atripla ([ATR]; the fixed-dose combination tablet containing FTC 200 mg/TDF 300 mg/EFV 600 mg) taken once daily until the end of the study (Week 240). At sites in France, the study was extended by a further 48 weeks (Year 6) or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.
  Interventions: Drug: Efavirenz (EFV); Drug: Lamivudine/zidovudine
- EFV+FTC+TDF (Experimental): Participants in this arm received 3 component drugs: efaviren (EFV; 600 mg) + emtricitabine (FTC; 200 mg) + tenofovir disoproxil fumarate (tenofovir DF [TDF]; 300 mg) as 3 separate pills once daily from the start of the study. At 96 weeks Truvada ([TVD] the fixed-dose combination pill containing FTC/TDF [200/300 mg] once daily) replaced the 2 component drugs FTC + TDF; participants continued to receive EFV 600 mg once daily. At Week 144 all participants who opted to roll over into the further 96-week study extension received ATR. At sites in France, the study was extended by a further 48 weeks (Year 6) or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.
  Interventions: Drug: Emtricitabine (FTC); Drug: Tenofovir Disoproxil Fumarate (TDF); Drug: Efavirenz (EFV); Drug: FTC/TDF; Drug: FTC/TDF/EFV

INTERVENTIONS:
Drug: Emtricitabine (FTC) — Capsule containing 200 mg FTC, taken once daily, for 96 weeks
  Other Names: Emtriva
  Arms: EFV+FTC+TDF
Drug: Tenofovir Disoproxil Fumarate (TDF) — Tablet containing 300 mg TDF, taken once daily, for 96 weeks
  Other Names: Viread
  Arms: EFV+FTC+TDF
Drug: Efavirenz (EFV) — Tablet containing 600 mg EFV, taken once daily, for 96 weeks
  Other Names: Sustiva
Drug: FTC/TDF — Fixed-dose combination tablet containing FTC 200 mg/TDF 300 mg, once daily, from Week 96 to 144
  Other Names: Truvada (TVD)
  Arms: EFV+FTC+TDF
Drug: FTC/TDF/EFV — Fixed-dose combination tablet containing FTC 200 mg/TDF 300 mg/EFV 600 mg, taken once daily, from Week 144 to 240
  Other Names: Atripla (ATR)
  Arms: EFV+FTC+TDF
Drug: Lamivudine/zidovudine — Fixed-dose combination tablet containing lamivudine 150 mg/zidovudine 300 mg, taken twice daily, for 240 weeks
  Other Names: Combivir (CBV)
  Arms: EFV+CBV

SUMMARY:
The purpose of Study GS-01-934 was to assess the efficacy and safety of two simplified antiretroviral treatment (ART) regimens in ART-naive, human immunodeficiency virus, type 1 (HIV-1) infected participants. The primary objective of the study was to assess noninferiority of emtricitabine (FTC) and tenofovir disoproxil fumarate (tenofovir DF; TDF) in combination with efavirenz (EFV) relative to Combivir (CBV) in combination with EFV in the treatment of HIV-1 infected ART-naive participants, determined by the achievement and maintenance of confirmed HIV-1 ribonucleic acid (RNA) < 400 copies/mL (c/mL) through Week 48, as defined by the United States (US) Food and Drug Administration (FDA) time-to-loss-of-virologic-response (TLOVR) algorithm.

DETAILED DESCRIPTION:
This study was originally planned as a 48-week, Phase 3, randomized, open-label, multicenter study comparing EFV+FTC+TDF (administered as the individual component drugs) versus CBV (lamivudine/zidovudine) + EFV to assess the efficacy and safety of both treatments in ART-Naive, HIV-1 infected participants. The regimen of CBV (administered twice daily) + EFV (administered once daily) served as the active control treatment and was compared with the regimen of EFV+FTC+TDF; each component drug in the EFV+FTC+TDF regimen was administered once daily.

Week 48 to Week 96:

The study was extended and continued to evaluate the efficacy and safety of the two regimens up to a total treatment duration of 96 weeks. The regimen of EFV+FTC+TDF continued to be dosed as the component drugs (EFV + FTC + TDF), once daily, without regard to meals. The regimen of CBV+EFV was dosed as 2 pills (CBV, twice daily in the morning without regard to meals) + EFV (once daily, without regard to meals).

Week 96 to Week 144:

A further study extension changed the 3-pill EFV+FTC+TDF regimen to a 2-pill regimen of EFV + Truvada ([TVD]: a fixed-dose combination pill containing FTC/TDF), once daily without regard to meals, and continued to evaluate the efficacy and safety of the two regimens for a further 48 weeks up to a total study treatment duration of 144 weeks. The regimen of CBV+EFV continued to be dosed as 2 pills (CBV, twice daily in the morning without regard to meals) + EFV (once daily, without regard to meals).

Week 144 to end of study (Week 240):

A final study extension provided all study participants from both treatment regimens the option to switch their respective treatments to the 1-pill regimen of for a further 96 weeks up to a total study duration of 240 weeks (5 years) to further assess the efficacy and safety of ART regimen simplification. At sites in France, the study was extended by a further 48 weeks (Year 6) or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.

ELIGIBILITY:
Inclusion Criteria: Participants must have met all inclusion criteria within 28 days prior to randomization unless specified otherwise including:

* Plasma HIV-1 RNA levels greater than 10,000 c/mL using Roche Amplicor HIV-1 Monitor Test Version 1.5 Standard
* Adequate renal function: Calculated creatinine clearance greater than or equal to 50 mL/min according to the Cockcroft-Gault Formula.
* Hepatic transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) 3 x upper limit of normal (ULN).
* Total bilirubin less than or equal to 1.5 mg/dL.
* Adequate hematologic function (absolute neutrophil count greater than or equal to 1,000/mm^3; platelets greater than or equal to 50,000/mm^3; hemoglobin greater than or equal to 8.0 g/dL).
* Serum amylase less than or equal to 1.5 x ULN.
* Serum phosphorus greater than or equal to 2.2 mg/dL.
* Willingness to use effective contraception by both males and females while on study treatment and for 30 days following study drug completion.
* Life expectancy greater than or equal to 1 year
* The ability to understand and sign written informed consent form obtained prior to initiation of study procedures.

Exclusion Criteria: Participants were not eligible for entry to the study if any of the following were met:

* Prior treatment with any non-nucleoside reverse transcriptase inhibitor (NNRTI), nucleoside reverse transcriptase inhibitor (NRTI), or protease inhibitor (PI).
* A new AIDS-defining condition diagnosed (exception CD4 criteria) within 30 days of baseline.
* Receiving ongoing therapy with any of the following: nephrotoxic agents, probenecid, systemic chemotherapeutic agents, systemic corticosteroids, interleukin-2, drugs that interact with efavirenz. Administration of any of the above medications must be discontinued at least 30 days prior to baseline visit and for duration of study.
* Pregnant or lactating participants.
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Participants with biopsy-confirmed KS were eligible but must not have received any systemic therapy for KS within 30 days of baseline and not anticipated starting systemic therapy during the study.
* Prior history of renal or bone disease.
* Any other clinical condition prior to therapy that would make the participant unsuitable for the study or unable to comply with the dosing requirements in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2003-07; Primary Completion 2005-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cheng, MD, PhD, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - AIDS Healthcare Foundation Research, Beverly Hills, California
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Orlando Immunology Center, Orlando, Florida
  - NorthStar Medical Center, Chicago, Illinois
  - Jemsek Clinic, Huntersville, North Carolina

REFERENCES:
- [Result] Gallant JE, DeJesus E, Arribas JR, Pozniak AL, Gazzard B, Campo RE, Lu B, McColl D, Chuck S, Enejosa J, Toole JJ, Cheng AK; Study 934 Group. Tenofovir DF, emtricitabine, and efavirenz vs. zidovudine, lamivudine, and efavirenz for HIV. N Engl J Med. 2006 Jan 19;354(3):251-60. doi: 10.1056/NEJMoa051871. PMID 16421366
- See also: Gilead Website — http://www.Gilead.com
- See also: Viread website — http://www.Viread.com
- See also: Sustiva website — http://www.Sustiva.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-01-934_144_wk_synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 70 study sites in the United States and Europe. The first participant was screened on 29 July 2003; the last participant was randomized on 16 January 2004; the last participant observation for the primary endpoint analysis was 11 February 2005; the last participant last visit for end of study analysis was 10 June 2009.
Pre-assignment Details: Of the 517 enrolled participants, 6 received no study drug (the safety analysis set was therefore 511 participants: 257 [efavirenz+emtricitabine+tenofovir disoproxil fumarate group] and 254 [efavirenz+combivir group], respectively).
Groups:
- EFV+FTC+TDF: Participants in this group received 3 component drugs: efavirenz (EFV) 600 mg + emtricitabine (FTC) 200 mg + tenofovir disoproxil fumarate (tenofovir DF; TDF) 300 mg, each once daily, from the start of the study. At 96 weeks Truvada ([TVD] the fixed-dose combination pill containing FTC/TDF (200 mg/300 mg) replaced FTC + TDF; participants continued to receive EFV as before. Nevirapine 200 mg twice daily could replace EFV in the event of efavirenz-associated central nervous system (CNS) toxicity.
  At Week 144 all participants who opted to roll over into the further 96-week study extension received Atripla ([ATR]; the fixed dose combination pill containing EFV/FTC/TDF, 600 mg/200 mg/300 mg) until the end of the study (Week 240). At sites in France, the study was extended by a further 48 weeks or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.
- CBV+EFV: Participants in this group received EFV 600 mg once daily + Combivir ([CBV]; the fixed dose combination pill containing lamivudine + zidovudine [150 mg/300 mg]) twice daily from the start of the study until Week 144. Nevirapine 200 mg twice daily could replace EFV in the event of efavirenz-associated CNS toxicity.
  At Week 144 all participants who opted to roll over into the additional 96-week study extension received ATR until the end of the study (Week 240). At sites in France, the study was extended by a further 48 weeks or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.
Period: Randomized Phase
Arm/Group | EFV+FTC+TDF | CBV+EFV
Started | 257 (Intention to treat (ITT) population N=255 (2 participants had received prior antiretroviral therapy)) | 254 (ITT analysis population)
Completed | 187 | 166
Not Completed | 70 | 88
Not completed — Lost to Follow-up | 26 | 33
Not completed — Adverse Event | 10 | 10
Not completed — Withrawal of consent | 10 | 18
Not completed — Sub-optimal virological response | 3 | 13
Not completed — Noncompliance | 8 | 4
Not completed — Protocol Violation | 2 | 0
Not completed — Pregnancy | 3 | 1
Not completed — Death | 1 | 3
Not completed — Hepatitis C treatment contraindicated | 0 | 1
Not completed — Inability to swallow pills | 0 | 1
Not completed — Incarceration | 3 | 2
Not completed — Moved out of State | 0 | 1
Not completed — Baseline NNRTI resistance mutations | 4 | 0
Not completed — High Hepatitis B DNA | 0 | 1
Period: Atripla Phase
Arm/Group | EFV+FTC+TDF | CBV+EFV
Started | 160 (Number of participants who completed randomized phase and opted to roll over to Atripla at Week 144) | 126 (Number of participants who completed randomized phase and opted to roll over to Atripla at Week 144)
Completed | 142 | 106
Not Completed | 18 | 20
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 5 | 7
Not completed — Pregnancy | 0 | 1
Not completed — Death | 0 | 2
Not completed — Withdrew consent | 7 | 7
Not completed — Sub-optimal virological response | 0 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EFV+FTC+TDF | CBV+EFV | Total
Number analyzed (Participants) | 255 | 254 | 509
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (9.9) | 38 (9.0) | 38 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 219 | 221 | 440
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 142 | 156 | 298
  Black | 65 | 51 | 116
  Hispanic | 39 | 40 | 79
  Asian | 3 | 3 | 6
  Not allowed to report | 0 | 1 | 1
  Other | 6 | 3 | 9
HIV Status [Number; unit: Participants]
  Asymptomatic | 33 | 26 | 59
  Symptomatic HIV Infection | 117 | 127 | 244
  AIDS | 105 | 101 | 206
CD4 cell count [Mean (Standard Deviation); unit: Cells/mm^3] | 246 (171.9) | 245 (156.6) | 245 (164.2)
HIV-1 RNA [Mean (Standard Deviation); unit: Log10 c/mL] | 5.03 (0.54) | 5.00 (0.51) | 5.01 (0.52)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 400 c/mL at Week 48 (Defined by the Food and Drug Administration [FDA] Time-to-Loss-of Virologic Response [TLOVR] Algorithm
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 400 c/mL had to satisfy the following criteria: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug except nevirapine in place of EFV prior to Week 48 visit; 2) achieved confirmed HIV-1 RNA < 400 c/mL on 2 consecutive visits prior to Week 48 visit (ie, the first of the 2 consecutive HIV-1 RNA < 400 c/mL occurred prior to the Week 48 visit; 3) not had confirmed HIV-1 RNA > 400 c/mL after achievement of confirmed HIV RNA levels < 400 c/mL prior to Week 48 visit.
Time Frame: 48 weeks
Population: Modified intention to treat (MITT) analysis set included all randomized participants who received at least 1 dose of study treatment, no major protocol violations, and no baseline primary NNRTI resistance mutation (2 participants were not ART-naive at study start; 22 participants had NNRTI resistance mutations at baseline [MITT analysis set: 487])
Measure: Number; unit: Percentage of participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of participants | 84.4 | 72.8
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: the percentage of responders (who achieved and maintained confirmed HIV-1 RNA < 400 c/mL [defined by the TLOVR algorithm]) through Week 48 in the EFV+FTC+TDF group is more than 13% worse than in the CBV+EFV group. Alternative Hypothesis: the percentage of responders who achieved and maintained confirmed HIV-1 RNA < 400 c/mL [defined by the TLOVR algorithm]) through Week 48 in the EFV+FTC+TDF group is no more than 13% worse than in the CBV+EFV group; Test type: Non-Inferiority or Equivalence — Assuming 70% response rate for each group at Week 48, 500 participants (250 per group) were sufficient to achieve at least 85% power to establish non-inferiority between the 2 study groups with a delta of 13%. The definition of clinical non-inferiority used a 'delta' of 0.13 (response rate was expressed as a decimal-valued number between 0 and 1). The EFV+FTC+TDF group was declared non-inferior to the CBV+EFV group if the lower confidence bound was > -0.13; p = 0.002, Cochran-Mantel-Haenszel — The difference and 95% CI are stratum-weighted on baseline CD4 using normal approximation. The p-value for the superiority test is from the Cochran-Mantel-Haenzel test stratified on baseline CD4 cell count; No other adjustments were made; Difference in percentages = 11.4, 95% CI 2-sided [4.3 to 18.6]

2. Secondary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 50 c/mL at Week 48 (Defined by FDA TLOVR Algorithm)
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 50 c/mL had to satisfy the following criteria: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug except nevirapine in place of EFV prior to Week 48 visit; 2) achieved confirmed HIV-1 RNA < 50 c/mL on 2 consecutive visits prior to Week 48 visit (that is, the first of the 2 consecutive HIV-1 RNA < 50 c/mL occurred prior to the Week 48 visit; 3) not had confirmed HIV-1 RNA > 50 c/mL after achievement of confirmed HIV RNA levels < 50 c/mL prior to Week 48 visit.
Time Frame: Week 48
Population: MITT analysis set included all randomized participants who received at least one dose of study medication, had no major protocol violations, and no baseline primary NNRTI resistance mutations (2 participants were not ART-naive at study start; 22 participants had NNRTI resistance mutations at baseline [MITT analysis set: 487])
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 79.5 | 70.4
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: the percentage of responders (who achieved and maintained confirmed HIV-1 RNA < 50 c/mL [defined by the TLOVR algorithm]) through Week 48 in the EFV+FTC+TDF group is more than 13% worse than in the CBV+EFV group. Alternative Hypothesis: the percentage of responders who achieved and maintained confirmed HIV-1 RNA < 50 c/mL [defined by the TLOVR algorithm]) through Week 48 in the EFV+FTC+TDF group is no more than 13% worse than in the CBV+EFV group; Test type: Non-Inferiority or Equivalence — The definition of clinical non-inferiority used a 'delta' of 0.13 (response rate was expressed as a decimal-valued number between 0 and 1). The EFV+FTC+TDF group was declared non-inferior to the CBV+EFV group if the lower confidence bound was > -0.13; p = 0.021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; No other adjustments were made; Difference in percentages = 9.1, 95% CI 2-sided [1.6 to 16.6]

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 400 c/mL at Week 48.
Description: The percentage of participants with plasma HIV-1 RNA < 400 c/mL at Week 48. Participants with missing observations/changes in ART were considered to have HIV-1 RNA ≥ 400 c/mL (i.e., ITT missing or switch=failure analysis).
Time Frame: 48 weeks
Population: Intention to Treat (ITT) analysis set (Missing Observation or Switch in ART=Failure). ITT analysis set included all randomized participants who received at least one dose of study medication, and had no major protocol violations (2 participants were not ART-naive at study start [ITT analysis set: 509]).
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of Participants | 80.4 | 69.3
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null hypothesis: The percentage of participants with HIV-1 RNA < 400 c/mL at Week 48 in the EFV+FTC+TDF group is more than 13% worse than the CBV+EFV group. Alternative hypothesis: The percentage of participants with HIV-1 RNA < 400 c/mL at Week 48 in the EFV+FTC+TDF group is no more than 13% worse than the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; No other adjustments were made; Difference in percentages = 11.2, 95% CI 2-sided [3.7 to 18.6]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 c/mL at Week 48
Description: The percentage of participants with plasma HIV-1 RNA < 50 c/mL at Week 48. Participants with missing observations/changes in ART were considered to have HIV-1 RNA ≥ 50 c/mL (i.e., ITT missing or switch=failure analysis).
Time Frame: 48 Weeks
Population: ITT analysis set (Missing Observation or Switch in ART=Failure). ITT analysis set included all randomized participants who received at least one dose of study medication, and had no major protocol violations (2 participants were not ART-naive at study start [ITT analysis set: 509]).
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of Participants | 74.5 | 66.9
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null hypothesis: The percentage of participants with HIV-1 RNA < 50 c/mL at Week 48 in the EFV+FTC+TDF group is more than 13% worse than the CBV+EFV group. Alternative hypothesis: The percentage of participants with HIV-1 RNA < 50 c/mL at Week 48 in the EFV+FTC+TDF group is no more than 13% worse than the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.058, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; No other adjustments were made; Difference in percentages = 7.9, 95% CI 2-sided [0.1 to 15.6]

5. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 400 c/mL) at Week 48
Description: TLOVR for participants who achieved a confirmed virologic response was the time to the earliest of: premature study regimen discontinuation or the first of 2 consecutive HIV-1 RNA ≥ 400 c/mL or last HIV-1 RNA ≥ 400 c/mL followed by loss to follow-up. If the time to HIV-1 RNA ≥ 400 c/mL was immediately preceded by missing scheduled visits then the time of virologic failure was replaced by the first such missing visit. Participants who had not achieved a confirmed virologic response before regimen discontinuation were considered "non-responders" on Study Day 1.
Time Frame: Baseline to 48 weeks
Population: ITT analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of Participants | 19 | 30
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with Loss of Virologic Response through Week 48 is equal between the two treatment groups. Alternative hypothesis: The percentage of participants with Loss of Virologic Response through Week 48 is different between the two treatment groups; Test type: Superiority or Other; p = 0.003, Log Rank — The distribution of time to loss-of-virologic response was estimated using the Kaplan-Meier product limit method and compared between treatment groups using a baseline CD4 stratum-weighted log-rank test; No other adjustments were made

6. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 50 c/mL) at Week 48
Description: TLOVR for participants who achieved a confirmed virologic response was the time to the earliest of: premature study regimen discontinuation or the first of 2 consecutive HIV-1 RNA ≥ 50 c/mL or last HIV-1 RNA ≥ 50 c/mL followed by loss to follow-up. If the time to HIV-1 RNA ≥ 50 c/mL was immediately preceded by missing scheduled visits then the time of virologic failure was replaced by the first such missing visit. Participants who had not achieved a confirmed virologic response before regimen discontinuation were considered "non-responders" on Study Day 1.
Time Frame: Baseline to 48 Weeks
Population: ITT analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of Participants | 23 | 32
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.046, Log Rank — [p-value comment as in outcome 5, analysis 1]; No other adjustments were made

7. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA < 400 c/mL) at Week 48
Description: Participants who achieved confirmed HIV-1 RNA < 400 c/mL but had not experienced a confirmed relapse were considered censored at the last HIV-1 RNA collection date.
Time Frame: Baseline to 48 Weeks
Population: ITT analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of Participants | 9 | 16
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 400 c/mL) at Week 48 is equal for the 2 treatment groups. Alternative Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 400 c/mL) at Week 48 is different between the 2 treatment groups; Test type: Superiority or Other; p = 0.026, Log Rank — The distribution of pure virological failure was estimated using the Kaplan-Meier product limit method and compared between treatment groups using a baseline CD4 stratum-weighted log-rank test; No other adjustments were made

8. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA < 50 c/mL) at Week 48
Description: Participants who achieved confirmed HIV-1 RNA < 50 c/mL but had not experienced a confirmed relapse were considered censored at the last HIV-1 RNA collection date.
Time Frame: Baseline to 48 Weeks
Population: ITT analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of participants | 16 | 24
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 50 c/mL) through Week 48 for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 50 c/mL) through Week 48 for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.063, Log Rank — [p-value comment as in outcome 7, analysis 1]; No other adjustments were made

9. Secondary Outcome: Change From Study Baseline in HIV-1 RNA (Log10 c/mL) at Week 48
Description: Change from study baseline to Week 48 in HIV-1 RNA in log10 scale (Week 48 HIV-1 RNA value in log10 scale minus study baseline HIV-1 RNA value in log10 scale).
Time Frame: Study baseline to Week 48
Population: As treated (AT) analysis set included all participants who received at least one dose of study medication and had not committed any major protocol violation.
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 201 | 172
Log10 c/mL | -3.31 (0.54) | -3.26 (0.58)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from baseline through Week 48 in plasma HIV-1 RNA for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from baseline through Week 48 in plasma HIV-1 RNA for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.31, Van Elteren — The change from baseline to Week 48 in HIV-1 RNA was compared between the 2 treatment groups using baseline CD4 stratum-weighted CI around the mean difference. P-value is from stratum-weighted Van Elteren test; No other adjustments were made; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.16 to 0.06]

10. Secondary Outcome: Change From Study Baseline in CD4 Cell Count (Cells/mm^3) at Week 48
Description: Change from study baseline to Week 48 in CD4 cell count = Week 48 CD4 cell count value minus study baseline CD4 cell count value
Time Frame: Study baseline to Week 48
Population: AT analysis set included all participants who received at least one dose of study medication and had not committed any major protocol violation.
Measure: Mean (Standard Deviation); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 199 | 164
CD4 Cell Count (cells/mm^3) | 190 (111.7) | 158 (107.3)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from baseline through Week 48 in CD4 cell count for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from baseline through Week 48 in CD4 cell count for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.002, Van Elteren — The change from baseline to Week 48 in HIV-1 RNA was compared between the 2 treatment groups using baseline CD4 stratum-weighted CI around the mean difference. P-value is from stratum weighted Van Elteren test; No other adjustments were made; stratum-weighted difference = 31.74, 95% CI [8.96 to 54.52]

11. Secondary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 400 c/mL at Week 96 (Defined by FDA TLOVR Algorithm)
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 400 c/mL had to satisfy the following criteria: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug except nevirapine in place of EFV prior to Week 96 visit; 2) achieved confirmed HIV-1 RNA < 400 c/mL on 2 consecutive visits prior to Week 96 visit (that is, the first of the 2 consecutive HIV-1 RNA < 400 c/mL occurred prior to the Week 96 visit; 3) not had confirmed HIV-1 RNA > 400 c/mL after achievement of confirmed HIV RNA levels < 400 c/mL prior to Week 96 visit.
Time Frame: 96 Weeks
Population: Week 96 efficacy analysis set excludes Week 48 responders who did not consent after Week 48 visits from MITT analysis set (Week 96 efficacy analysis set: [463])
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 232 | 231
Percentage of Participants | 74.6 | 61.9
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: the percentage of responders (who achieved and maintained confirmed HIV-1 RNA < 400 c/mL [defined by the TLOVR algorithm]) through Week 96 in the EFV+FTC+TDF group is more than 13% worse than in the CBV+EFV group. Alternative Hypothesis: the percentage of responders who achieved and maintained confirmed HIV-1 RNA < 400 c/mL [defined by the TLOVR algorithm]) through Week 96 in the EFV+FTC+TDF group is no more than 13% worse than in the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.004, Cochran-Mantel-Haenszel — The difference and 95% CI are stratum weighted on baseline CD4 using normal approximation. The p-value for the superiority test is from Cochran-Mantel-Haenszel test stratified on baseline CD4 cell count; No other adjustments were made; Difference in percentages = 12.7, 95% CI 2-sided [4.3 to 21.1]

12. Secondary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 50 c/mL at Week 96 (Defined by FDA TLOVR Algorithm)
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 50 c/mL had to satisfy the following criteria: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug except nevirapine in place of EFV prior to Week 96 visit; 2) achieved confirmed HIV-1 RNA < 50 c/mL on 2 consecutive visits prior to Week 96 visit (that is, the first of the 2 consecutive HIV-1 RNA < 50 c/mL occurred prior to the Week 96 visit; 3) not had confirmed HIV-1 RNA > 50 c/mL after achievement of confirmed HIV RNA levels < 50 c/mL prior to Week 96 visit.
Time Frame: Week 96
Population: Week 96 efficacy analysis excludes Week 48 responders who did not consent after Week 48 visits from MITT analysis set (Week 96 efficacy analysis set: [465])
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 232 | 233
Percentage of Participants | 67.2 | 60.9
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: the percentage of responders (who achieved and maintained confirmed HIV-1 RNA < 50 c/mL [defined by the TLOVR algorithm]) through Week 96 in the EFV+FTC+TDF group is more than 13% worse than in the CBV+EFV group. Alternative Hypothesis: the percentage of responders who achieved and maintained confirmed HIV-1 RNA < 50 c/mL [defined by the TLOVR algorithm]) through Week 96 in the EFV+FTC+TDF group is no more than 13% worse than in the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.158, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; No other adjustments were made; Difference in proportions = 6.4, 95% CI 2-sided [-2.3 to 15.0]

13. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 400 c/mL) at Week 96
Description: TLOVR for participants with confirmed virologic response (2 consecutive HIV-1 RNA < 400 c/mL) prior to study drug discontinuation, was the time to the earliest of premature study regimen discontinuation, or confirmed HIV-1 RNA > 400 c/mL (2 consecutive HIV-1 RNA ≥ 400 c/mL, or the last HIV-1 RNA ≥ 400 c/mL followed by premature study regimen discontinuation due to loss to follow-up). Participants who did not achieve confirmed virologic response before premature study regimen discontinuation or last HIV-1 RNA, were assumed to have lost virologic response on Study Day 1.
Time Frame: Week 96
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 25 | 37
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Ther percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 400 c/mL) at Week 96 for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative Hypothesis: The percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 400 c/mL) at Week 96 for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.003, Log Rank — [p-value comment as in outcome 5, analysis 1]; No other adjustments were made

14. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 50 c/mL) at Week 96
Description: as for outcome 6
Time Frame: Week 96
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 32 | 38
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 50 c/mL) through Week 96 for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative Hypothesis: The percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 50 c/mL) through Week 96 for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.124, Log Rank — [p-value comment as in outcome 5, analysis 1]; No other adjustments were made

15. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA < 400 c/mL) at Week 96
Description: as for outcome 7
Time Frame: Week 96
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 9 | 17
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 400 c/mL) at Week 96 is equal for the 2 treatment groups. Alternative Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 400 c/mL) at Week 96 is different between the 2 treatment groups; Test type: Superiority or Other; p = 0.025, Log Rank — [p-value comment as in outcome 7, analysis 1]; No other adjustments were made

16. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA < 50 c/mL) at Week 96
Description: as for outcome 8
Time Frame: Week 96
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 20 | 23
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with pure virological failure (HIV-1 RNA < 50 c/mL) through Week 96 for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative Hypothesis: The percentage of participants with pure virological failure (HIV-1 RNA < 50 c/mL) through Week 96 for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.41, Log Rank — [p-value comment as in outcome 7, analysis 1]; No other adjustments were made

17. Secondary Outcome: Change From Study Baseline in HIV-1 RNA (Log10 c/mL) at Week 96
Description: Change from study baseline to Week 96 in HIV-1 RNA in log10 scale (Week 96 HIV-1 RNA value in log10 scale minus study baseline HIV-1 RNA value in log10 scale).
Time Frame: Study baseline to Week 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 170 | 145
Log10 c/mL | -3.30 (0.57) | -3.25 (0.59)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from baseline through Week 96 in plasma HIV-1 RNA for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from baseline through Week 96 in plasma HIV-1 RNA for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.45, Van Elteren — The change from baseline to Week 96 in HIV-1 RNA was compared between the 2 treatment groups using baseline CD4 stratum-weighted CI around the mean difference; No other adjustments were made; stratum-weighted difference = -0.05, 95% CI [-0.17 to 0.08]

18. Secondary Outcome: Change From Study Baseline in CD4 Cell Count (Cells/mm^3) at Week 96
Description: Change from study baseline to Week 96 in CD4 cell count = Week 96 CD4 cell count value minus study baseline CD4 cell count value
Time Frame: Baseline to Week 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 166 | 142
CD4 Cell Count (cells/mm^3) | 270 (147.5) | 237 (136.4)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from baseline through Week 96 in CD4 cell count for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from baseline through Week 96 in CD4 cell count for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.036, Van Elteren — The change from baseline to Week 96 in CD4 cell count was compared between the 2 treatment groups using baseline CD4 stratum-weighted CI around the mean difference. P-value is from stratum weighted Van Elteren test; No other adjustments were made; stratum-weighted difference = 32.93, 95% CI [0.87 to 64.99]

19. Secondary Outcome: Change in Limb Fat (kg) From Week 48 to Week 96
Description: Change from Week 48 to Week 96 in limb fat = Week 96 limb fat value minus Week 48 limb fat value.
Time Frame: Week 48 to Week 96
Population: ITT (whole body dual-energy X-ray absorptiometry [DEXA] scans to determine limb fat content were conducted only at selected sites at Week 48 and Week 96. ITT analysis set: 93)
Measure: Mean (Standard Deviation); unit: limb fat (kg)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 49 | 44
limb fat (kg) | 0.74 (1.60) | -0.77 (1.58)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Change from Week 48 to Week 96 in limb fat for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Change from Week 48 to Week 96 in limb fat for the EFV+FTC+TDF and CBV+EFV groups are not equal; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The change from Week 48 to Week 96 in limb fat was compared between the 2 treatment groups; the P-value is from the Wilcoxon Rank Sum Test; No other adjustments were made

20. Secondary Outcome: Change in Trunk Fat (kg) From Week 48 to Week 96
Description: Change from Week 48 to Week 96 in trunk fat = Week 96 trunk fat value minus Week 48 trunk fat value
Time Frame: Week 48 to Week 96
Population: ITT (whole body DEXA scans to determine trunk fat content were conducted only at selected sites at Week 48 and Week 96. ITT analysis set: 93)
Measure: Mean (Standard Deviation); unit: trunk fat (kg)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 49 | 44
trunk fat (kg) | 0.94 (2.30) | -0.04 (1.65)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from Week 48 to Week 96 in Trunk Fat for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from Week 48 to Week 96 in Trunk Fat for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.025, Wilcoxon Rank Sum test — The change from Week 48 to Week 96 in trunk fat was compared between the 2 treatment groups; the P-value is from the Wilcoxon Rank Sum Test; No other adjustments were made

21. Secondary Outcome: Change in Total Body Fat (kg) From Week 48 to Week 96
Description: Change from Week 48 to Week 96 in total body fat = Week 96 total body fat value minus Week 48 total body fat value
Time Frame: 48 weeks to 96 weeks
Population: ITT (whole body DEXA scans to determine total body fat content were conducted only at selected sites at Week 48 and Week 96. ITT analysis set for limb fat analyses: 93)
Measure: Mean (Standard Deviation); unit: total body fat (kg)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 49 | 44
total body fat (kg) | 1.69 (3.80) | -0.82 (3.01)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from Week 48 to Week 96 in Total Body Fat for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from Week 48 to Week 96 in Total Body Fat for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum test — [p-value comment as in outcome 20, analysis 1]; No other adjustments were made

22. Secondary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 400 c/mL at Week 144 (Defined by FDA TLOVR Algorithm)
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 400 c/mL had to satisfy the following: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug, except nevirapine in place of EFV, prior to Week 144 visit; 2) achieved confirmed HIV-1 RNA < 400 c/mL on 2 consecutive visits prior to Week 144 visit (i.e., the first of the 2 consecutive HIV-1 RNA < 400 c/mL occurred prior to the Week 144 visit; 3) not had confirmed HIV-1 RNA > 400 c/mL after achievement of confirmed HIV-1 RNA levels < 400 c/mL prior to Week 144 visit.
Time Frame: 144 weeks
Population: Week 144 Efficacy Analysis set (excludes the Week 96 responders who did not consent after Week 96 visits from Week 96 efficacy analysis set [Week 144 efficacy analysis set: 456).
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 227 | 229
Percentage of Participants | 70.9 | 58.1
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: the proportion of responders (who achieved and maintained confirmed HIV-1 RNA < 400 c/mL [defined by the TLOVR algorithm]) through Week 144 in the EFV+FTC+TDF group is more than 13% worse than in the CBV+EFV group. Alternative Hypothesis: the proportion of responders who achieved and maintained confirmed HIV-1 RNA < 400 c/mL [defined by the TLOVR algorithm]) through Week 144 in the EFV+FTC+TDF group is no more than 13% worse than in the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.004, Cochran-Mantel-Haenszel — The difference and 95% CI are stratum weighted on baseline CD4 using normal approximation. The p-value for the superiority test is from Cochran-Mantel-Haenzel test; No other adjustments were made; Difference in proportions = 12.9, 95% CI 2-sided [4.2 to 21.6]

23. Secondary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 50 c/mL at Week 144 (Defined by FDA TLOVR Algorithm)
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 50 c/mL (c/mL) had to satisfy the following criteria: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug, except nevirapine in place of EFV, prior to Week 144 visit; 2) achieved confirmed HIV-1 RNA < 50 c/mL on 2 consecutive visits prior to Week 144 visit (that is, the first of the 2 consecutive HIV-1 RNA < 50 c/mL occurred prior to the Week 144 visit; 3) not had confirmed HIV-1 RNA > 50 c/mL after achievement of confirmed HIV-1 RNA levels < 50 c/mL prior to Week 144 visit.
Time Frame: Week 144
Population: Week 144 Efficacy Analysis set (excludes the Week 96 responders who did not consent after Week 96 visits from Week 96 efficacy analysis set [Week 144 efficacy analysis set: 458).
Measure: Number; unit: Percentage of participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 227 | 231
Percentage of participants | 64.3 | 56.3
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: the proportion of responders (who achieved and maintained confirmed HIV-1 RNA < 50 c/mL [defined by the TLOVR algorithm]) through Week 144 in the EFV+FTC+TDF group is more than 13% worse than in the CBV+EFV group. Alternative Hypothesis: the proportion of responders who achieved and maintained confirmed HIV-1 RNA < 50 c/mL [defined by the TLOVR algorithm]) through Week 144 in the EFV+FTC+TDF group is no more than 13% worse than in the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.082, Cochran-Mantel-Haenszel — The difference and 95% CI are stratum weighted on baseline CD4 using normal approximation. The p-value for the superiority test is from the Cochran-Mantel-Haenszel test stratified on baseline CD4 cell count; No other adjustments were made; Difference in proportions = 8.1, 95% CI 2-sided [-0.8 to 17.0]

24. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 400 c/mL at Week 144
Description: The percentage of participants with plasma HIV-1 RNA < 400 c/mL at Week 144. Participants with missing observations/changes in ART were considered to have HIV-1 RNA ≥ 400 c/mL (i.e., ITT missing or switch=failure analysis).
Time Frame: Week 144
Population: ITT Analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of Participants | 63.1 | 51.6
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with HIV-1 RNA < 400 c/mL at Week 144 in the EFV+FTC+TDF group is more than 13% worse than the CBV+EFV group. Alternative hypothesis: The percentage of participants with HIV-1 RNA < 400 c/mL at Week 144 in the EFV+FTC+TDF group is no more than 13% worse than the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.009, Cochran-Mantel-Haenszel — The difference and 95% CI are stratum weighted on baseline CD4 using normal approximation. The p-value for the superiority test is from Cochran-Mantel-Haenzel test stratified on baseline CD4 cell count; No other adjustments were made; Difference in proportions = 11.6, 95% CI [3.1 to 20.1]

25. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 50 c/mL at Week 144
Description: The percentage of participants with plasma HIV-1 RNA < 50 c/mL at Week 144. Participants with missing observations/changes in ART were considered to have HIV-1 RNA ≥ 50 c/mL (i.e., ITT missing or switch=failure analysis).
Time Frame: Week 144
Population: ITT Analysis set (Missing Observation or Switch in ART=Failure)
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 255 | 254
Percentage of Participants | 60.8 | 50.4
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null hypothesis: The percentage of participants with HIV-1 RNA < 50 c/mL at Week 144 in the EFV+FTC+TDF group is more than 13% worse than the CBV+EFV group. Alternative hypothesis: The percentage of participants with HIV-1 RNA < 50 c/mL at Week 144 in the EFV+FTC+TDF group is no more than 13% worse than the CBV+EFV group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.019, Cochran-Mantel-Haenszel — The p-value for the superiority test is from Cochran-Mantel-Haenzel test stratified on baseline CD4 cell count; No other adjustments were made; Difference in proportions = 10.4, 95% CI 2-sided [1.8 to 19.0]

26. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 400 c/mL) at Week 144
Description: as for outcome 5
Time Frame: Week 144
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 28 | 41
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 400 c/mL) through Week 144 for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative Hypothesis: The percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 400 c/mL) through Week 144 for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.003, Log Rank — The distribution of loss of virological response was estimated using the Kaplan-Meier product limit method and compared between treatment groups using a baseline CD4 stratum-weighted log-rank test; No other adjustments were made

27. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 50 c/mL) at Week 144
Description: as for outcome 6
Time Frame: Week 144
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 34 | 43
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 50 c/mL) through Week 144 for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative Hypothesis: The percentage of participants with loss of virologic response (confirmed HIV-1 RNA < 50 c/mL) through Week 144 for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.056, Log Rank — [p-value comment as in outcome 7, analysis 1]; No other adjustments were made

28. Secondary Outcome: Percentage of Participants With Pure Virological Failure (HIV-1 RNA < 400 c/mL) at Week 144
Description: as for outcome 7
Time Frame: Week 144
Population: MITT
Measure: Number; unit: Percentage of participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of participants | 11 | 17
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 400 c/mL) at Week 144 is equal for the 2 treatment groups. Alternative Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 400 c/mL) at Week 144 is different between the 2 treatment groups; Test type: Superiority or Other; p = 0.066, Log Rank — [p-value comment as in outcome 7, analysis 1]; No other adjustments were made

29. Secondary Outcome: Percentage of Participants With Pure Virological Failure (HIV-1 RNA < 50 c/mL) at Week 144
Description: as for outcome 8
Time Frame: Week 144
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 244 | 243
Percentage of Participants | 21 | 25
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 50 c/mL) at Week 144 is equal for the 2 treatment groups. Alternative Hypothesis: The percentage of participants with pure virological failure (confirmed HIV-1 RNA < 50 c/mL) at Week 144 is different between the 2 treatment groups; Test type: Superiority or Other; p = 0.30, Log Rank — [p-value comment as in outcome 7, analysis 1]; No other adjustments were made

30. Secondary Outcome: Change From Study Baseline in HIV-1 RNA (Log10 c/mL) at Week 144
Description: Change from study baseline to Week 144 in HIV-1 RNA in log10 scale (Week 144 HIV-1 RNA value in log10 scale minus study baseline HIV-1 RNA value in log10 scale).
Time Frame: Study baseline to Week 144
Population: AT analysis set
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 160 | 124
Log10 c/mL | -3.32 (0.54) | -3.30 (0.52)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from baseline to Week 144 in plasma HIV-1 RNA for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from baseline to Week 144 in plasma HIV-1 RNA for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.39, Van Elteren — The change from baseline to Week 144 in HIV-1 RNA was compared between the 2 treatment groups using baseline CD4 stratum-weighted CI around the mean difference. P-value is from a stratum weighted Van Elteren test; No other adjustments were made; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.16 to 0.08]

31. Secondary Outcome: Change From Study Baseline in CD4 Cell Count (Cells/mm^3) at Week 144
Description: Change from study baseline to Week 144 in CD4 cell count = Week 144 CD4 cell count value minus study baseline CD4 cell count value
Time Frame: Baseline to Week 144
Population: AT analysis set
Measure: Mean (Standard Deviation); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 152 | 122
CD4 Cell Count (cells/mm^3) | 312 (161.2) | 271 (147.4)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from baseline toWeek 144 in CD4 cell count for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from baseline to Week 144 in CD4 cell count for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.089, Van Elteren — The change from baseline to Week 144 in CD4 cell count was compared between the 2 treatment groups using baseline CD4 stratum-weighted CI around the mean difference. P-value is from a stratum weighted Van Elteren test; No other adjustments were made; Mean Difference (Net) = 41.30, 95% CI 2-sided [4.05 to 78.55]

32. Secondary Outcome: Change in Limb Fat (kg) From Week 48 to Week 144
Description: Change from Week 48 to Week 144 in limb fat = Week 144 limb fat value minus Week 48 limb fat value
Time Frame: Week 48 to Week 144
Population: ITT (whole body DEXA scans to determine limb fat content were conducted only at selected sites at Week 48, Week 96 and Week 144. ITT analysis set: 86)
Measure: Mean (Standard Deviation); unit: limb fat (kg)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 48 | 38
limb fat (kg) | 1.13 (1.93) | -1.09 (1.72)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from Week 48 baseline to Week 144 in Limb Fat for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from Week 48 baseline to Week 144 in Limb Fat for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.001, Wilcoxon Rank Sum test — P-value is from the Wilcoxon Rank Sum Test; No other adjustments were made

33. Secondary Outcome: Change in Trunk Fat (kg) From Week 48 to Week 144
Description: Change from Week 48 to Week 144 in trunk fat = Week 144 trunk fat value minus Week 48 trunk fat value
Time Frame: Week 48 to Week 144
Population: ITT (whole body DEXA scans to determine trunk fat content were conducted only at selected sites at Week 48, Week 96 and Week 144. ITT analysis set: 86)
Measure: Mean (Standard Deviation); unit: trunk fat (kg)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 48 | 38
trunk fat (kg) | 1.30 (2.40) | -0.10 (1.79)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from Week 48 baseline to Week 144 in Trunk Fat for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from Week 48 baseline to Week 144 in Trunk Fat for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p = 0.011, Wilcoxon Rank Sum test — P-value is from the Wilcoxon Rank Sum Test; No other adjustments were made

34. Secondary Outcome: Change in Total Body Fat (kg) From Week 48 to Week 144
Description: Change from Week 48 to Week 144 in total body fat = Week 144 total body fat value minus Week 48 total body fat value
Time Frame: Week 48 to Week 144
Population: ITT (whole body DEXA scans to determine total body fat content were conducted only at selected sites at Week 48, Week 96 and Week 144. ITT analysis set: 86)
Measure: Mean (Standard Deviation); unit: total body fat (kg)
Arm/Group | EFV+FTC+TDF | CBV+EFV
Number analyzed (Participants) | 48 | 38
total body fat (kg) | 2.47 (4.22) | -1.18 (3.37)
Statistical Analysis 1: Comparison: EFV+FTC+TDF vs CBV+EFV; Null Hypothesis: Changes from Week 48 baseline to Week 144 in Total Body Fat for the EFV+FTC+TDF and CBV+EFV groups are equal. Alternative hypothesis: Changes from Week 48 baseline to Week 144 in Total Body Fat for the EFV+FTC+TDF and CBV+EFV groups are different; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum test — P-value is from the Wilcoxon Rank Sum Test; No other adjustments were made

35. Secondary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 400 c/mL at Week 240 (Atripla Week 96) Defined by the FDA TLOVR Algorithm
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 400 c/mL had to satisfy the following criteria: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug except nevirapine in place of EFV prior to Week 240 visit; 2) achieved confirmed HIV-1 RNA < 400 c/mL on 2 consecutive visits prior to Week 240 visit (that is, the first of the 2 consecutive HIV-1 RNA < 400 c/mL occurred prior to the Week 240 visit; 3) not had confirmed HIV-1 RNA > 400 c/mL after achievement of confirmed HIV RNA levels < 400 c/mL prior to Week 240 visit.
Time Frame: Week 144 (Atripla baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set (all participants who received at least one dose of Atripla). Data collected after permanent discontinuation of the study regimen was excluded from this analysis set.
Measure: Number; unit: Percentage of Participants
Groups:
- All Atripla: Participants rolled over into the 96-week study extension and received Atripla ([ATR]; the fixed dose combination pill containing EFV/FTC/TDF) until the end of the study (Week 240). At sites in France, the study was extended by a further 48 weeks (Year 6) or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.
Arm/Group | All Atripla
Number analyzed (Participants) | 286
Percentage of Participants | 87

36. Secondary Outcome: Percentage of Participants With Confirmed Plasma HIV-1 RNA < 50 c/mL at Week 240 (Atripla Week 96) Defined by the FDA TLOVR Algorithm
Description: Participants who achieved/maintained confirmed HIV-1 RNA < 50 c/mL had to satisfy the following criteria: 1) not experienced death, permanent study drug discontinuation, or addition of new antiretroviral drug except nevirapine in place of EFV prior to Week 240 visit; 2) achieved confirmed HIV-1 RNA < 50 c/mL on 2 consecutive visits prior to Week 240 visit (that is, the first of the 2 consecutive HIV-1 RNA < 50 c/mL occurred prior to the Week 240 visit; 3) not had confirmed HIV-1 RNA > 50 c/mL after achievement of confirmed HIV RNA levels < 50 c/mL prior to Week 240 visit.
Time Frame: Week 144 (Atripla baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 286
Percentage of Participants | 85

37. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 400 c/mL at Week 240 (Atripla Week 96)
Description: The percentage of participants with plasma HIV-1 RNA < 400 c/mL at Week 240. Participants with missing observations/changes in ART were considered to have HIV-1 RNA ≥ 400 c/mL (i.e., ITT missing or switch=failure analysis).
Time Frame: Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Percentage of Participants
Groups:
- EFV+FTC+TDF/Atripla (From Study Baseline): Participants in this group were originally randomized to receive the 3 component drugs: efavirenz (EFV) + emtricitabine (FTC) + tenofovir disoproxil fumarate (tenofovir DF; TDF) for 96 weeks, and subsequently received Truvada ([TVD] the fixed-dose combination pill containing FTC/TDF) and EFV until Week 144. Participants then rolled over into the further 96-week study extension and received Atripla ([ATR]; the fixed dose combination pill containing EFV/FTC/TDF) until the end of the study (Week 240). At sites in France, the study was extended by a further 48 weeks (Year 6) or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.
- All Atripla (From Atripla Baseline): Participants rolled over into the 96-week study extension and received Atripla ([ATR]; the fixed dose combination pill containing EFV/FTC/TDF) until the end of the study (Week 240). At sites in France, the study was extended by a further 48 weeks (Year 6) or until ATR became commercially available (whichever happened first); once ATR became commercially available in France participants were not required to complete the full 288 weeks of the study.
Arm/Group | EFV+FTC+TDF/Atripla (From Study Baseline) | All Atripla (From Atripla Baseline)
Number analyzed (Participants) | 160 | 286
Percentage of Participants | 87 | 85

38. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 50 c/mL at Week 240 (Atripla Week 96)
Description: The percentage of participants with plasma HIV-1 RNA < 50 c/mL at Week 240. Participants with missing observations/changes in ART were considered to have HIV-1 RNA ≥ 50 c/mL (i.e., ITT missing or switch=failure analysis).
Time Frame: Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF/Atripla (From Study Baseline) | All Atripla (From Atripla Baseline)
Number analyzed (Participants) | 160 | 286
Percentage of Participants | 84 | 82

39. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 400 c/mL) From Week 144 (Atripla Baseline) Through Week 240 (Atripla Week 96)
Description: as for outcome 5
Time Frame: Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 286
Percentage of Participants | 13

40. Secondary Outcome: Percentage of Participants With Loss of Virologic Response (HIV-1 RNA < 50 c/mL) From Week 144 (Atripla Baseline) Through Week 240 (Atripla Week 96)
Description: as for outcome 6
Time Frame: Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 286
Percentage of Participants | 15

41. Secondary Outcome: Percentage of Participants With Pure Virological Failure (HIV-1 RNA < 400 c/mL) Through Week 240 (Atripla Week 96)
Description: as for outcome 7
Time Frame: Week 240 (Atripla Week 96)
Population: MITT Analysis Set (EFV+FTC+TDF group from study baseline; N=244).
  Atripla Efficacy Analysis Set (All Atripla Group from Atripla baseline; N=286)
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF/Atripla (From Study Baseline) | All Atripla (From Atripla Baseline)
Number analyzed (Participants) | 244 | 286
Percentage of Participants | 11 | 2

42. Secondary Outcome: Percentage of Participants With Pure Virological Failure (HIV-1 RNA < 50 c/mL) Through Week 240 (Atripla Week 96)
Description: as for outcome 8
Time Frame: Week 240 (Atripla Week 96)
Population: as for outcome 41
Measure: Number; unit: Percentage of Participants
Arm/Group | EFV+FTC+TDF/Atripla (From Study Baseline) | All Atripla (From Atripla Baseline)
Number analyzed (Participants) | 244 | 286
Percentage of Participants | 22 | 4

43. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at Week 240 (Atripla Week 96)
Description: Change from baseline to Week 240 (Atripla Week 96) in CD4 cell count = Week 240 (Atripla Week 96) CD4 cell count value minus baseline CD4 cell count value
Time Frame: Study/Atripla baseline to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: CD4 Cell count (Cells/mm^3)
Arm/Group | EFV+FTC+TDF/Atripla (From Study Baseline) | All Atripla (From Atripla Baseline)
Number analyzed (Participants) | 138 | 243
CD4 Cell count (Cells/mm^3) | 346 (197.2) | 42 (148.2)

44. Secondary Outcome: Change in Limb Fat (kg) From Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Description: Change from Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96) in limb fat = Week 240 (Atripla Week 96) limb fat value minus Week 144 (Atripla Baseline) limb fat value
Time Frame: Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: limb fat (kg)
Arm/Group | All Atripla
Number analyzed (Participants) | 213
limb fat (kg) | 0.12 (1.657)
Statistical Analysis 1: Comparison: All Atripla; Null Hypothesis: Change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) limb fat value is equal to zero. Alternative hypothesis: Change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) limb fat value is not equal to zero; Test type: Superiority or Other; p = 0.16, Wilcoxon Signed Rank test — P-value is from the Wilcoxon Signed Rank test. No adjustments for multiple comparisons were made

45. Secondary Outcome: Change in Trunk Fat (kg) From Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Description: Change from Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96) in trunk fat = Week 240 (Atripla Week 96) trunk fat value minus Week 144 (Atripla Baseline) trunk fat value
Time Frame: Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: trunk fat (kg)
Arm/Group | All Atripla
Number analyzed (Participants) | 213
trunk fat (kg) | 0.27 (2.242)
Statistical Analysis 1: Comparison: All Atripla; Null Hypothesis: Change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) trunk fat value is equal to zero. Alternative hypothesis: Change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) trunk fat value is not equal to zero; Test type: Superiority or Other; p = 0.049, Wilcoxon Signed Rank test — P-value is from the Wilcoxon Signed Rank test. No adjustments for multiple comparisons were made

46. Secondary Outcome: Change in Total Body Fat (kg) From Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Description: Change from Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96) in total body fat = Week 240 (Atripla Week 96) total body fat value minus Week 144 (Atripla Baseline) total body fat value
Time Frame: Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: total body fat (kg)
Arm/Group | All Atripla
Number analyzed (Participants) | 212
total body fat (kg) | 0.37 (3.747)
Statistical Analysis 1: Comparison: All Atripla; Null Hypothesis: Change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) total body fat value is equal to zero. Alternative hypothesis: Change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) total body fat value is not equal to zero; Test type: Superiority or Other; p = 0.055, Wilcoxon Signed Rank test — P-value is from the Wilcoxon Signed Rank test. No adjustments for multiple comparisons were made

47. Secondary Outcome: Treatment Satisfaction Questionnaire (Satisfaction With Convenience and Simplicity of Current Treatment Regimen): Change From Week 144 to Week 240 in the Category Shift From Atripla Baseline.
Description: Participants were asked: "In general, how satisfied are you with the convenience and simplicity of your current treatment regimen?" Possible responses were on a 4-category scale: "very satisfied"; "somewhat satisfied"; "somewhat dissatisfied"; and "very dissatisfied". For the evaluation of changes in treatment satisfaction from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) responses were dichotomized into "very satisfied" and "not very satisfied" ("not very satisfied" included "very dissatisfied"; "somewhat dissatisfied"; and "somewhat satisfied").
Time Frame: Week 144 ([W 144]; Atripla baseline) to Week 240 ([W 240]; Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 225
Participants
  Very satisfied (W 144 and W 240) | 182
  Not very satisfied (W 144 and W 240) | 6
  Very satisfied (W 144); not very satisfied (W 240) | 8
  Not very satisfied (W 144); very satisfied (W 240) | 29
Statistical Analysis 1: Comparison: All Atripla; Null Hypothesis: There is no category shift from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96). Alternative Hypothesis: There is a category shift from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96); Test type: Superiority or Other; p < 0.001, McNemar — The number and proportion of participants in each category ("very satisfied", "not very satisfied") were summarized. The P-value for the category shift from Week 144 baseline within a treatment group was calculated using the McNemar test

48. Secondary Outcome: Treatment Satisfaction Questionnaire (Satisfaction With Current Treatment Regimen to Control HIV): Change From Week 144 to Week 240 in the Category Shift From Atripla Baseline.
Description: Participants were asked: "In general, how satisfied are you with the ability of your current treatment regimen to control your HIV infection?" Possible responses were on a 4-category scale: "very satisfied"; "somewhat satisfied"; "somewhat dissatisfied"; and "very dissatisfied". For the evaluation of changes in treatment satisfaction from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) responses were dichotomized into "very satisfied" and "not very satisfied" ("not very satisfied" included "very dissatisfied"; "somewhat dissatisfied"; and "somewhat satisfied").
Time Frame: Week 144 ([W 144]; Atripla baseline) to Week 240 ([W 240]; Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 226
Participants
  Very satisfied (W 144 and W 240) | 192
  Not very satisfied (W 144 and W 240) | 8
  Very satisfied (W 144); not very satisfied (W 240) | 9
  Not very satisfied (W 144); very satisfied (W 240) | 17
Statistical Analysis 1: Comparison: All Atripla; [analysis description as in outcome 47, analysis 1]; Test type: Superiority or Other; p = 0.12, McNemar — [p-value comment as in outcome 47, analysis 1]

49. Secondary Outcome: Treatment Satisfaction Questionnaire (Satisfaction With Tolerability of Current Treatment Regimen) Change From Week 144 to Week 240 in the Category Shift From Atripla Baseline.
Description: Participants were asked: "In general, how satisfied are you with your ability to tolerate your current treatment regimen?" Possible responses were on a 4-category scale: "very satisfied"; "somewhat satisfied"; "somewhat dissatisfied"; and "very dissatisfied". For the evaluation of changes in treatment satisfaction from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) responses were dichotomized into "very satisfied" and "not very satisfied" ("not very satisfied" included "very dissatisfied"; "somewhat dissatisfied"; and "somewhat satisfied").
Time Frame: Week 144 ([W 144]; Atripla baseline) to Week 240 ([W 240]; Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 226
Participants
  Very satisfied (W 144 and W 240) | 166
  Not very satisfied (W 144 and W 240) | 21
  Very satisfied (W 144); not very satisfied (W 240) | 13
  Not very satisfied (W 144); very satisfied (W 240) | 26
Statistical Analysis 1: Comparison: All Atripla; [analysis description as in outcome 47, analysis 1]; Test type: Superiority or Other; p = 0.037, McNemar — [p-value comment as in outcome 47, analysis 1]

50. Secondary Outcome: Treatment Satisfaction Questionnaire (General Satisfaction With Current Treatment Regimen): Change From Week 144 to Week 240 in the Category Shift From Atripla Baseline.
Description: Participants were asked: "In general, how satisfied are you with your current treatment regimen?" Possible responses were on a 4-category scale: "very satisfied"; "somewhat satisfied"; "somewhat dissatisfied"; and "very dissatisfied". For the evaluation of changes in treatment satisfaction from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) responses were dichotomized into "very satisfied" and "not very satisfied" ("not very satisfied" included "very dissatisfied"; "somewhat dissatisfied"; and "somewhat satisfied").
Time Frame: Week 144 ([W 144]; Atripla baseline) to Week 240 ([W 240]; Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 222
Participants
  Very satisfied (W 144 and W 240) | 180
  Not very satisfied (W 144 and W 240) | 10
  Very satisfied (W 144); not very satisfied (W 240) | 9
  Not very satisfied (W 144); very satisfied (W 240) | 23
Statistical Analysis 1: Comparison: All Atripla; [analysis description as in outcome 47, analysis 1]; Test type: Superiority or Other; p = 0.013, McNemar — [p-value comment as in outcome 47, analysis 1]

51. Secondary Outcome: Treatment Satisfaction Questionnaire (Bothered With the Side Effects of Current Treatment Regimen): Change From Week 144 to Week 240 in the Category Shift From Atripla Baseline.
Description: Participants were asked: "How bothered are you with the side effects of your current treatment regimen?" Possible responses were on a 4-category scale: "does not bother me"; "bothers me a little bit"; "bothers me a lot"; and "bothers me terribly". For the evaluation of the change in treatment satisfaction from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) responses were dichotomized into "does not bother me" and "bothers me" ("bothers me" included "bothers me a little bit"; "bothers me a lot"; "bothers me terribly").
Time Frame: Week 144 ([W 144]; Atripla baseline) to Week 240 ([W 240]; Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Number; unit: Participants
Arm/Group | All Atripla
Number analyzed (Participants) | 226
Participants
  Bothers me (W 144 and W 240) | 41
  Does not bother me (W 144 and W 240) | 126
  Bothers me (W 144); does not bother me (W 240) | 31
  Does not bother me (W 144); bothers me (W 240) | 28
Statistical Analysis 1: Comparison: All Atripla; [analysis description as in outcome 47, analysis 1]; Test type: Superiority or Other; p = 0.70, McNemar — The number and proportion of participants in each category ("bothers", "does not bother") were summarized. The P-value for the category shift from Week 144 baseline within a treatment group was calculated using the McNemar test

52. Secondary Outcome: Quality of Life (SF-12v2 Health Survey: Physical Component Summary) Change From Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Description: The change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) in the SF-12v2 Health Survey: Physical Component Summary (PCS). The SF-12v2 includes 8 concepts commonly represented in health surveys: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. Results are expressed in terms of 2 composite scores: the PCS and the Mental Component Summary (MCS). PCS and MCS values can range from 0 to 100 and are designed to have a mean value of 50 and SD of 10 (in the general population).
Time Frame: Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: Composite Score
Arm/Group | All Atripla
Number analyzed (Participants) | 213
Composite Score | 0.0 (6.80)
Statistical Analysis 1: Comparison: All Atripla; Null Hypothesis: There is no change in the PCS score from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96). Alternative Hypothesis: There is a change in the PCS score from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96); Test type: Superiority or Other; p = 0.95, Wilcoxon Signed Rank Test — P-value is from the Wilcoxon Signed Rank Test

53. Secondary Outcome: Quality of Life (SF-12v2 Health Survey: Mental Component Summary) Change From Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Description: The change from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96) in the SF-12v2 Health Survey MCS. The SF-12v2 includes 8 concepts commonly represented in health surveys: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. Results are expressed in terms of 2 composite scores: the PCS and the MCS. PCS and MCS values can range from 0 to 100 and are designed to have a mean value of 50 and a SD of 10 (in the general population).
Time Frame: Week 144 (Atripla Baseline) to Week 240 (Atripla Week 96)
Population: Atripla Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: Composite Score
Arm/Group | All Atripla
Number analyzed (Participants) | 213
Composite Score | 0.9 (8.65)
Statistical Analysis 1: Comparison: All Atripla; Null Hypothesis: There is no change in the MCS score from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96). Alternative Hypothesis: There is a change in the MCS score from Week 144 (Atripla baseline) to Week 240 (Atripla Week 96); Test type: Superiority or Other; p = 0.23, Wilcoxon Signed Rank Test — P-value is from the Wilcoxon Signed Rank Test

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported during the 144-week randomized treatment phase (FTC+TDF+EFV and CBV+EFV groups) and for the 96-week non-randomized Atripla extension phase (for all participants who opted to switch to Atripla).
Description: AEs are reported for the FTC+TDF+EFV and CBV+EFV groups from baseline through to Week 144 and for all participants who opted to receive ATR from Week 144 to 240 (All Atripla group). AEs are also reported for those participants who received FTC+TDF+EFV from baseline until Week 144 and opted to receive ATR until Week 240/288 (FTC+TDF+EFV/ATR group).
Groups:
- FTC+TDF+EFV (Baseline to 144 Weeks): Exposure to the component drugs EFV+FTC+TDF during the randomized treatment phase was up to 144 weeks (TVD replaced FTC+TDF from Week 96). For this safety population, N=257.
- FTC+TDF+EFV/ATR (Baseline to 240 Weeks): Exposure to the component drugs EFV+FTC+TDF during the randomized treatment phase and during the Atripla treatment phase was up to 240 weeks (TVD replaced FTC+TDF at Week 96; ATR replaced TVD+EFV at Week 144). Exposure to ATR for 6 participants at sites in France was up to 288 weeks (this was due to a protocol amendment which allowed these participants to continue to receive ATR until it became commercially available). For this safety population, N=160.
- CBV+EFV (Baseline to 144 Weeks): Exposure to CBV+EFV during the randomized treatment phase was up to 144 weeks. For this safety population, N=254.
- All Atripla (Week 144 to 240): Exposure for all participants from both treatment groups who switched to ATR at Week 144 and continued treatment to Week 240 was up to 96 weeks. Exposure to ATR for 6 participants at sites in France was up to 144 weeks (this was due to a protocol amendment which allowed these participants to continue to receive ATR until it became commercially available). For this safety population, N=286.
Arm/Group | FTC+TDF+EFV (Baseline to 144 Weeks) | FTC+TDF+EFV/ATR (Baseline to 240 Weeks) | CBV+EFV (Baseline to 144 Weeks) | All Atripla (Week 144 to 240)
Serious Adverse Events (participants affected / at risk) | 29/257 | 24/160 | 35/254 | 14/286
Other Adverse Events (participants affected / at risk) | 233/257 | 152/160 | 222/254 | 190/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC+TDF+EFV (Baseline to 144 Weeks) (N=257) | FTC+TDF+EFV/ATR (Baseline to 240 Weeks) (N=160) | CBV+EFV (Baseline to 144 Weeks) (N=254) | All Atripla (Week 144 to 240) (N=286)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 7 | 0
Anal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 2 | 2 | 2 | 0
Basedow's Disease (Endocrine disorders) | 1 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Cardiac Disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Catheter Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis Staphylococcus (Infections and infestations) | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 1
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia Bacteriemia (Infections and infestations) | 0 | 0 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroenteritis Cryptosporidial (Infections and infestations) | 1 | 1 | 0 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypercreatinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Immune Reconstitution Syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis Cryptococcal (Infections and infestations) | 1 | 0 | 1 | 0
Meningitis Viral (Infections and infestations) | 0 | 0 | 1 | 0
Meningorrhagia (Nervous system disorders) | 1 | 1 | 0 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Mycobacterium Avium Complex Infection (Infections and infestations) | 0 | 0 | 1 | 0
Mycobacterium Kansasii Infection (Infections and infestations) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 2 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Nodal Rhythm (Cardiac disorders) | 1 | 1 | 0 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peripheral Ischemia (Vascular disorders) | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 2 | 1
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 0 | 0 | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Rectal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Secondary Syphilis (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Splenectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Staphylococcal Abscess (Infections and infestations) | 0 | 0 | 2 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 2 | 0 | 2
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Tonsillitis Streptococcal (Infections and infestations) | 1 | 1 | 0 | 0
Transient Ischemic Attack (Nervous system disorders) | 1 | 1 | 0 | 0
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC+TDF+EFV (Baseline to 144 Weeks) (N=257) | FTC+TDF+EFV/ATR (Baseline to 240 Weeks) (N=160) | CBV+EFV (Baseline to 144 Weeks) (N=254) | All Atripla (Week 144 to 240) (N=286)
Abdominal Pain (Gastrointestinal disorders) | 12 | 9 | 14 | 4
Abnormal Dreams (Psychiatric disorders) | 45 | 33 | 34 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 17 | 0
Anogenital Warts (Infections and infestations) | 10 | 9 | 14 | 5
Anxiety (Psychiatric disorders) | 15 | 15 | 19 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 17 | 14 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 26 | 24 | 20 | 16
Bronchitis (Infections and infestations) | 22 | 21 | 14 | 9
Chest Pain (General disorders) | 0 | 8 | 0 | 3
Conjunctivitis (Eye disorders) | 0 | 13 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 32 | 31 | 15
Depression (Psychiatric disorders) | 38 | 30 | 32 | 21
Diarrhoea (Gastrointestinal disorders) | 73 | 57 | 50 | 29
Dizziness (Nervous system disorders) | 71 | 50 | 74 | 9
Dyspepsia (Gastrointestinal disorders) | 8 | 8 | 15 | 5
Ear Infection (Infections and infestations) | 0 | 9 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 10 | 0 | 3
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 9 | 0 | 2
Fatigue (General disorders) | 46 | 34 | 46 | 14
Folliculitis (Infections and infestations) | 15 | 12 | 12 | 2
Gastroenteritis (Infections and infestations) | 0 | 9 | 0 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 8 | 0 | 4
Haemorrhoids (Gastrointestinal disorders) | 10 | 11 | 13 | 7
Headache (Nervous system disorders) | 51 | 40 | 43 | 16
Herpes Simplex (Infections and infestations) | 18 | 0 | 21 | 0
Herpes Zoster (Infections and infestations) | 12 | 13 | 13 | 8
Hypertension (Vascular disorders) | 0 | 13 | 0 | 11
Influenza (Infections and infestations) | 19 | 17 | 11 | 12
Insomnia (Psychiatric disorders) | 44 | 38 | 45 | 22
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 8 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 13 | 11 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 16 | 9 | 11
Nasopharyngitis (Infections and infestations) | 45 | 49 | 33 | 42
Nausea (Gastrointestinal disorders) | 66 | 37 | 83 | 6
Night Sweats (Skin and subcutaneous tissue disorders) | 16 | 9 | 9 | 6
Onychomycosis (Infections and infestations) | 0 | 13 | 0 | 5
Oral Herpes (Infections and infestations) | 0 | 10 | 0 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 0 | 8
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 12 | 0 | 7
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 0 | 28 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 16 | 12 | 15 | 4
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 0 | 5
Pyrexia (General disorders) | 24 | 24 | 17 | 12
Rash (Skin and subcutaneous tissue disorders) | 39 | 27 | 33 | 8
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 0 | 3
Seasonal Allergy (Immune system disorders) | 0 | 18 | 0 | 12
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 21 | 12
Sinusitis (Infections and infestations) | 33 | 35 | 17 | 19
Somnolence (Nervous system disorders) | 18 | 12 | 17 | 0
Syphilis (Infections and infestations) | 0 | 11 | 0 | 11
Tinea Pedis (Infections and infestations) | 0 | 10 | 0 | 8
Tooth Abscess (Infections and infestations) | 0 | 9 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 48 | 49 | 27 | 30
Vomiting (Gastrointestinal disorders) | 20 | 15 | 33 | 3
Weight Decreased (Investigations) | 0 | 9 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may publish study results 2 years after the completion of the study or earlier with the advance written permission of Gilead. The PI will submit any proposed publication or presentation of study results together with the name of the proposed scientific journal, forum or confeence to Gilead prior to submission or presentation (30 days prior for manuscripts and 15 days for abstracts and oral presentations).